CLINICAL TRIAL: NCT01576874
Title: The Gender-Sex Hormone Interface With Craving & Stress-Related Changes in Smoking
Acronym: SCOR-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Gray, MD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Kevin Gray, MD, Professor, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00016931; P50DA016511 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Nicotine Dependence
Keywords: nicotine dependence; hormones
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxytocin (Experimental): Participants will be administered 40 IUs of oxytocin nasal spray at one study visit.
  Interventions: Drug: Oxytocin
- placebo (Placebo Comparator): Participants will be administered 40 IUs of placebo nasal spray at one study visit.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Oxytocin — 40 IUs of oxytocin administered intranasally one time
  Other Names: syntocinon
  Arms: oxytocin
Drug: placebo — placebo administered intranasally one time
  Arms: placebo

SUMMARY:
The purpose of the overall parent study is to determine the impact of gender and hormones (estradiol, progesterone, testosterone and cortisol) on responses to stress and smoking cues presented in daily, "real-world" cue presentations compared to a final cue session in a lab. In addition, in the portion of the study that incorporates clinical trials elements and is reported here, the study will examine the impact of a single dose of oxytocin (chemical produced in the body) versus placebo (inactive substance) on reactivity to a stress procedure (Trier Social Stress Task) in smokers.

The overall parent study involves a cue presentation technology known as "CREMA" (Cue Reactivity Ecologic Momentary Assessment) which delivers four daily cue presentations to you on a handheld device during your everyday routine. Additionally, the study involves daily collection of saliva samples for hormonal testing. These daily procedures will provide information about the role of cues and hormones in daily life. The clinical trial portion of the study (reported here) consists of measures collected within the laboratory.

DETAILED DESCRIPTION:
Despite considerable advances in treatment development, cigarette smoking remains the leading cause of preventable death in the United States, and most smokers engaged in treatment are unsuccessful in quitting. The burden of illness is disproportionately borne by female smokers, who are less responsive to cessation interventions than males. The relationships between stress, craving, and smoking behavior are recognized as key factors underlying gender differences in nicotine dependence, but must be better understood and characterized to yield avenues for interventions addressing this critical health disparity.

In prior and ongoing SCOR studies, our research team has demonstrated gender and menstrual cycle/sex hormone influences on reactivity to laboratory-presented cues. Building from these laboratory findings, we propose taking two important next steps: (1) evaluating the experience of craving in the "real world" natural environment of female and male smokers, and (2) examining the impact of a safe and novel pharmacological intervention (oxytocin) on stress reactivity in female and male smokers.

If, as hypothesized, gender, sex hormones, and oxytocin administration influence the relationships between stress, craving, and smoking behavior, the findings could substantially address a key gender-related health disparity. Such knowledge could also inform the development of gender-specific interventions to enhance female smokers' response to cessation treatments. Therefore, the knowledge to be gained from the proposed study may yield significant public health benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males age 18 - 45 who smoke at least an average of 5 cigarettes per day for at least past 6 months
2. Females must be post menarche and pre-menopausal, have a regular menstrual cycle between 25 and 35 days, and, if recently pregnant, be at least three months post-delivery/breast feeding
3. Participants must submit a carbon monoxide sample of ≥ 5 ppm at their screening visit

Exclusion Criteria:

1. Any serious or unstable medical or psychiatric disorder that may, in the judgment of the study physician, interfere with study completion
2. Participants must not meet criteria for PTSD
3. Any medication (e.g., propranolol) that may interfere with psychophysiological (e.g., heart rate) monitoring
4. Current substance dependence other than nicotine and caffeine use, in the past month
5. Use of other tobacco products
6. Females must not be pregnant, breast feeding, status post hysterectomy or bilateral oophorectomy, or taking birth control or hormone replacement medication that would affect the menstrual cycle
7. Males must not be status post orchiectomy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2012-06; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saladin, PhD, Principal Investigator — Medical University of South Carolina; Kevin M Gray, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 72 | 72
Completed | 72 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 72 | 144
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (7.1) | 31.6 (7.7) | 31 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 27 | 26 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 28 | 54
  White | 41 | 40 | 81
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Craving Response to Trier Social Stress Task
Description: The TSST is the gold standard for evoking stress response in the laboratory. The participant must deliver a speech as though speaking to a group of hiring managers. The participant has 5 min to prepare, then three individuals unfamiliar to the participant (the audience) enter the room and are seated; the participant is instructed give the speech (without notes). The speech is delivered for 5 min, then the participant is instructed to serially subtract 13 from 1,022 as quickly and accurately as possible. The mental math recitation continues for 5 min, and at its conclusion, the spokesperson instructs the participant to stop and be seated, and the audience leaves the room. The total time for the TSST is 15 min.
  The Craving Questionnaire (Carter & Tiffany, 2001) is the sum of 4 items, each rated 1-5 on a Likert scale, with total score ranging 4-20, and higher scores indicating higher craving.
Time Frame: Immediately after the conclusion of the TSST
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 72 | 72
units on a scale | 16.18 (4.78) | 16.69 (4.78)

2. Secondary Outcome: Stress Response to Trier Social Stress Task
Description: The TSST is the gold standard for evoking stress response in the laboratory. The participant must deliver a speech as though speaking to a group of hiring managers. The participant has 5 min to prepare, then three individuals unfamiliar to the participant (the audience) enter the room and are seated; the participant is instructed give the speech (without notes). The speech is delivered for 5 min, then the participant is instructed to serially subtract 13 from 1,022 as quickly and accurately as possible. The mental math recitation continues for 5 min, and at its conclusion, the spokesperson instructs the participant to stop and be seated, and the audience leaves the room. The total time for the TSST is 15 min.
  The single stress item is derived from the CREMA Mood/Stress Assessment (Warthen & Tiffany, 2009), asking how stressed the participant felt at that time, on a 5-point Likert scale, ranging 1-5 with higher score indicating feeling more stressed
Time Frame: Immediately after the conclusion of the TSST
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 72 | 72
units on a scale | 2.81 (1.43) | 2.57 (1.23)

3. Secondary Outcome: Cortisol Response to Trier Social Stress Task
Description: Cortisol measured immediately following the Trier Social Stress Task, to evaluate physiological stress response.
Time Frame: Immediately following the Trier Social Stress Task
Measure: Mean (Standard Deviation); unit: micrograms per deciliter
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 72 | 72
micrograms per deciliter | 0.25 (0.13) | 0.25 (0.14)

ADVERSE EVENTS:
Time Frame: During laboratory visit after oxytocin or placebo administration (up to 3 hours after medication administration; any unresolved AEs at the end of the laboratory session are followed post-session to conclusion/resolution).
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT01576874/Prot_SAP_000.pdf